CLINICAL TRIAL: NCT06506708
Title: Effect of Massage and Hydrotherapy to Improve Well-being and Pain Perception in Women With Endometriosis Unresponsive to Conventional Treatment
Brief Title: Effect of Massage and Hydrotherapy to Improve Well-being and Pain Perception in Endometriosis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Francisco Artacho Cordón, Proffesor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAMMAM
Record Dates: First submitted 2024-07-03; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Endometriosis; Chronic Pelvic Pain Syndrome
MeSH Terms: conditions — Endometriosis | interventions — Hydrotherapy; Massage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care group (No Intervention): The gynecologist will proceed to administer the standard treatments to the control group. Moreover, assessors will emphasize healthy lifestyle benefits.
- Experimental group (Experimental): The comprehensive Hammam experience will consist of 3 sessions at the Arab baths of Hammam Al Ándalus, Granada -Spain- (once session each two weeks). Each session will involve a thermal circuit lasting approximately 75 minutes, following the institution's guidelines, inviting women to explore the warm, hot, and cold water baths, as well as the steam room. The thermal circuit will be complemented by a 15-minute relaxing Swedish massage using essential oils. During the final session, massage will be preceeded by a traditional Kessa treatment on a hot stone bed. During sessions, women will be involved in a multisensory experience, including aromatherapy and relaxing music, and where they will also have the opportunity to sipping on mint tea and relax on a building all decorated in resplendent Arabian décor. One member of the research team will be responsible for coordinating the sessions in collaboration with the Al Ándalus institution, subject to their availability.
  Interventions: Other: Hydrotherapy + massage

INTERVENTIONS:
Other: Hydrotherapy + massage — The comprehensive Hammam experience will consist of 3 sessions at the Arab baths of Hammam Al Ándalus, Granada -Spain- (once every two weeks). Each session will involve a thermal circuit lasting approximately 75 minutes, following the institution's guidelines, inviting women to explore the warm, hot, and cold water baths, as well as the steam room. The thermal circuit will be complemented by a 15-minute relaxing massage using essential oils. During the final session, massage will be preceeded by a traditional Kessa treatment on a hot stone bed. During sessions, women will be involved in a multisensory experience, including aromatherapy and where they will also have the opportunity to sipping on mint tea and relax on a building all decorated in resplendent Arabian décor. One member of the research team will be responsible for coordinating the sessions in collaboration with the Al Ándalus institution, subject to their availability.
  Arms: Experimental group

SUMMARY:
The objective is to analyze the short-term effect of a comprehensive HAMMAM experience combining therapeutic hydrotherapy, aromatherapy, music therapy, and Swedish massage on objective parameters and patient-reported outcomes related to well-being generation and pain reduction in women with endometriosis-related chronic pelvic pain.

DETAILED DESCRIPTION:
The main objective of this project is to analyze the short-term effect of a comprehensive HAMMAM experience combining therapeutic hydrotherapy, aromatherapy, music therapy, and Swedish massage on objective parameters and patient-reported outcomes related to well-being generation and pain reduction in women with endometriosis-related chronic pelvic pain (CPP).

For this purpose, a two-arm pre-post intervention study will be conducted, randomizing 44 women with CPP (22 in the intervention group and 22 in the control group). The intervention group, in addition to following the treatment proposed by their gynecologist, will participate in a comprehensive HAMMAM experience consisting of 3 sessions (one session each 14 days), where they will undergo a 75-minute thermal circuit (cold, warm and hot water pools) and a 15-minute of Swedish massage with a special focus in the abdomino-lumbo-pelvic region. During the last session, massage will be precceded by a 15-min traditional Kessa massage. During kessa massage, women will lie on a hot stone table for 15 minutes, while the skin is covered with red grape soap suds and scrubbed with a cotton fiber glove (kessa). The scrubbing will cleanse the skin of any dirt and residues, which may help them achieve a fully relaxed feeling

As participants in the intervention group, those in the the control group will receive the treatment stipulated by their gynecologist.

Participants will be evaluated before the start of the intervention (t0), and at the end of the last session (t1) on both self-reported variables (subjective well-being scale, satisfaction with life scale, quality of life, pain intensity, pain interference and pain catastrophizing scale), and objective variables (pressure pain thresholds).

Treatment efficacy will be analyzed using ANCOVA through SPSS v24.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic pain during the last 6 months more or equal to 4 in a NRS scale.
* Diagnosed with endometriosis (through surgery, magnetic resonance imaging or ultrasound imaging)
* Premenopausal status
* Be able to walk without assistance and to read and write enough
* Be capable and willing to provide consent

Exclusion Criteria:

* Acute or terminal illness
* A recent fracture in any upper or lower extremity (<3 months), disc herniation and any chronic disease or orthopaedic issues that would interfere with her ability to participate in this intervention program
* Express unwillingness to complete the study requirements
* Be involved in other rehabilitation program

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain intensity assessed by NRS | Baseline and immediately after intervention
  Numeric Rating Scale (NRS) will be used to identify self-reported levels of chronic pelvic pain, dysmenorrhea, dyspareunia, dyschezia and dysuria.. Scores range from 0 to 10. Higher scores represent increased pain intensity

SECONDARY OUTCOMES:
Changes in Pain Interference assessed by BPI | Baseline and immediately after intervention
  Brief Pain Inventory (BPI) will be used to address the interference of pain with daily life activities, scored in a 11-point Likert-type scale, where higher scores indicate higher pain interference.
Changes in Pressure pain threshold (PPT) assessed by algometry | Baseline and immediately after intervention
  Algometry will be used to measure PPT levels in abdomen, pelvis and lower back regions through an electronic algometer. For this purpose, an approximate rate of 0.3 kilograms/s will be applied with a 1cm2 probe. Seven points from the abdominal and pelvic area, and two additional points from the lower back region will be tested. Prior PPT assessment, assessor will ask for participants to press the switch when they first feel a change from pressure to pain. The mean of three tests, spaced by 30 s, will be used for the analysis.
Changes in Catastrophizing thoughts assessed by PCS | Baseline and immediately after intervention
  The Pain Catastrophizing Scale (PCS) will be also used to assess catastrophic thinking related to pain. Scores of this 13-item scale range from 0 to 52. Higher scores represent higher catastrophic thoughts.
Changes in quality of life assessed by EHP-30 | Baseline and immediately after intervention
  It will be assessed using the Endometriosis Health Profile-30 (EHP-30). It is a self-administered disease-specific instrument to measure QoL in women with endometriosis. The 30-item EHP, referred to the last 4 weeks, is comprised of five domains: pain, control and powerlessness, emotional well-being, social support, and self-image. Items within each subscale, answered on a 5-point Likert-type scale, are summed and then transformed to a percentage scale ranging from 0 (best health status) to 100 (worse health status) by dividing the raw score of all items by the maximum possible raw score, multiplied by 100
Changes in functioning assessed by PROMIS-29 | Baseline and immediately after intervention
  The Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) will be used. The PROMIS-29 is a 29-item instrument designed to measure functioning in a wide variety of clinical situations. It is divided in subscales (Physical Function; Anxiety; Depression; Fatigue; Sleep Disturbance; Ability to Participate in Social Roles and Activities; Pain Interference and Pain Intensity). Each item is scored from 1 to 5; a higher score indicates a higher degree of the construct being measured. For the subscales Physical Function and Ability to Participate in Social Roles and Activities, a higher score indicates better functioning, whereas for the other subscales a higher score indicates worse functioning.
Changes in Subjective well-being assessed by EBS-20 | Baseline and immediately after intervention
  The subjective Well-being Scale (EBS-20) will be used. This scale is comprised by 20 items, scored in a 6-point Likert-type scale. The mean score is calculated, with higher scores representing higher well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Artacho-Cordón, Principal Investigator — Universidad de Granada
Locations (1):
- Francisco Artacho Cordón, Granada, Spain

IPD SHARING:
Plan to Share IPD: No